CLINICAL TRIAL: NCT04795986
Title: First Clinical Evaluation of HEARO Robotic Cochlear Implantation Surgery in Austria
Acronym: HEARO-AT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Principal Investigator, Christoph Arnoldner, Assoc.-Prof. Priv.-Doz. Dr., Medical University of Vienna
Other Study IDs: HEARO-AT
Record Dates: First submitted 2021-02-22; First posted 2021-03-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Deafness
Keywords: cochlear implantation; robotic surgery; automated inner ear access; automated middle ear access
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: HEARO Procedure — robotic access to the middle and inner ear in cochlear implantation

SUMMARY:
To demonstrate the efficacy of a minimally invasive direct cochlear access via the HEARO procedure in cochlear implantation.

DETAILED DESCRIPTION:
The HEARO procedure involves a robot which drills the access to the cochlear in cochlear implantation.

The study is an observational study of the first implementation in clinical routine in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Adult cochlear implant candidates with suitable anatomy opting for a MED-EL cochlear implant.

Exclusion Criteria:

* Age under 18 years

  * Pregnant women
  * Facial recess size does not allow a minimum distance of 0.4mm from the planned trajectory to the facial nerve and 0.3mm to the chorda tympani
  * Vulnerable or mentally retarded candidates
  * Invalid or withdrawn informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cochlear implant candidates with suitable anatomy opting for a MED-EL cochlear implant.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of cochlear access | at implantation
  Percentage of patients with successful cochlear access with the hearo procedure (successful meaning no conventional mastoidectomy and posterior tympanotomy necessary)

SECONDARY OUTCOMES:
electrode array insertion outcomes | at implantation
  Percentage of patients with full electrode insertion (all contacts inside the cochlea) as assessed by postoperative DVT Imaging
Safety of cochlear access | at implantation
  Number of patients with facial nerve paralysis after cochlear implantation as assessed by the House-Brackmann scale.

CONTACTS AND LOCATIONS:
Locations (1):
- HNO Klinik am AKH Wien, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No